CLINICAL TRIAL: NCT01637792
Title: Randomized Controlled Trial Comparing Residual Kidney Function in Patients Undergoing Three or Four Exchanges CAPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Aiwu Lin, MD, PhD, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 044119620; 07QA14040 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality); 08DZ1900501 (Other Grant/Funding Number: Science and Technology Commission of Shanghai Municipality)
Record Dates: First submitted 2012-07-01; First posted 2012-07-11 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: End Stage Renal Disease; Anuria; Peritonitis
Keywords: peritoneal dialysis; dose; residual kidney function; technique survival; patient survival; peritonitis
MeSH Terms: conditions — Kidney Failure, Chronic; Anuria; Peritonitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Three 2-liter exchanges group (Experimental): A group of randomly assigned patients undergoing three 2-liter exchanges daily CAPD.
  Interventions: Other: Three 2-liter exchanges daily CAPD
- Four 2-liter exchanges group (Active Comparator): A group of randomly assigned patients undergoing four 2-liter exchanges daily CAPD.
  Interventions: Other: Four 2-liter exchanges daily CAPD

INTERVENTIONS:
Other: Three 2-liter exchanges daily CAPD — CAPD regimen of three 2-liter daily exchanges
  Other Names: small volume CAPD
  Arms: Three 2-liter exchanges group
Other: Four 2-liter exchanges daily CAPD — CAPD regimen of four 2-liter daily exchagnes
  Other Names: standard volume CAPD
  Arms: Four 2-liter exchanges group

SUMMARY:
The purpose of this study was to explore the impacts of different continuous ambulatory peritoneal dialysis (CAPD) dosage (three 2-Liter exchanges CAPD vs. four 2-Liter exchanges CAPD) on residual kidney function, technique survival, patient survival, and peritonitis in incident Chinese peritoneal dialysis patients.

DETAILED DESCRIPTION:
1. The primary end point for this study was changes in residual kidney function including GFR, daily urine volume (Uvol), and anuria-free survival. GFR and Uvol were evaluated within 1 week before CAPD initiation (the baseline), and then at month 1, 6, 12, 18 and 24. At the same time, body weight, blood pressure, daily net ultrafiltration, dialysis adequacy, peritoneal solute transport rate, and biochemical parameters etc. were assessed. Once an episode of peritonitis or other serious reversible intercurrent illness occurred, all the assessments were delayed one month after being cured. Anuria was termed by daily Uvol permanently less than 100 ml.
2. The secondary end points included technique survival, patient survival and peritonitis. Technique failure was defined as switching to maintenance hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

* incident CAPD patients aged 18 to 80 years
* GFR ≥ 2 ml/min and Uvol ≥ 500 ml/day

Exclusion Criteria:

* have a history of maintenance hemodialysis or renal transplantation
* anticipated life expectancy less than 6 months
* with active malignancy, acute infection, significant heart failure or in other severe conditions
* unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2004-06; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Residual kidney function including glomerular filtration rate (GFR), daily urine voume (Uvol), and anuria-free survival. | Up to 24 months after CAPD initiation
  GFR was calculated by the mean of renal clearance of urea and creatinine from a 24-h urine collection. Anuria was termed as consistently Uvol < 100 ml/day for more than a month.

SECONDARY OUTCOMES:
Number of participants having technique failure refering to switching to maintenance hemodialyisis | Up to 24 months after CAPD initiation.
Number of participants died | Up to 24 months after CAPD initiation
Episodes of peritonitis | Up to 24 months after CAPD initiation

CONTACTS AND LOCATIONS:
Overall Officials: Wei Fang, MD, PhD, Principal Investigator — Renal Division, Renji Hospital, Shanghai Jiaotong University School of Medicine
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lo WK, Jiang Y, Cheng SW, Cheng IK. Survival of CAPD patients in a center using three two-liter exchanges as standard regime. Perit Dial Int. 1996;16 Suppl 1:S163-6. PMID 8728185
- [Background] Szeto CC, Lai KN, Yu AW, Leung CB, Ho KK, Mak TW, Li PK, Lam CW. Dialysis adequacy of Asian patients receiving small volume continuous ambulatory peritoneal dialysis. Int J Artif Organs. 1997 Aug;20(8):428-35. PMID 9323505
- [Background] Fang W, Qian J, Lin A, Rowaie F, Ni Z, Yao Q, Bargman JM, Oreopoulos DG. Comparison of peritoneal dialysis practice patterns and outcomes between a Canadian and a Chinese centre. Nephrol Dial Transplant. 2008 Dec;23(12):4021-8. doi: 10.1093/ndt/gfn372. Epub 2008 Sep 12. PMID 18790809
- [Background] Singhal MK, Bhaskaran S, Vidgen E, Bargman JM, Vas SI, Oreopoulos DG. Rate of decline of residual renal function in patients on continuous peritoneal dialysis and factors affecting it. Perit Dial Int. 2000 Jul-Aug;20(4):429-38. PMID 11007375